CLINICAL TRIAL: NCT03672006
Title: Tissue Plasminogen Activator Dwells to Reduce Catheter-associated Thrombosis and Infection
Brief Title: t-PA Prophylaxis to Prevent Catheter-associated Thrombosis and Infection
Acronym: TOPCAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Sheila Hanson, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MCWisconsin
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Central Venous Catheter Thrombosis; Central Venous Catheter Associated Bloodstream Infection
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis | interventions — Tissue Plasminogen Activator; Tetradecanoylphorbol Acetate; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Centralized pharmacy will prepare and blind the study drug (t-PA) and the control (heparin)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- alteplase (Experimental): patients will receive 30 min-4 hours dwells of alteplase (recombinant t-PA) (2mg/2ml, up to 2mg per dose) to central venous catheter every 3 days (maximum 10 doses)
  Interventions: Biological: alteplase (recombinant t-PA)
- Heparin (Active Comparator): patients will receive 30 min-4 hours heparin (10U/ml, up to 2 ml per dose) dwells to central venous catheter every 3 days (maximum 10 doses)
  Interventions: Drug: Heparin

INTERVENTIONS:
Biological: alteplase (recombinant t-PA) — Medication administered to dwell in central venous catheter
  Other Names: tpa
  Arms: alteplase
Drug: Heparin — Medication administered to dwell in central venous catheter
  Other Names: control
  Arms: Heparin

SUMMARY:
The purpose of this pilot study is to test feasibility of concept, consent and enrollment rates, and mechanics of study designed to assess if intra-catheter dwells of tissue plasminogen activator (t-PA) is effective in decreasing the rate of clinically diagnosed central line associated blood stream infection (CLABSI) or venous thromboembolism (VTE) in central venous catheters (CVC) compared to standard of care heparin dwell.

DETAILED DESCRIPTION:
This pilot study Children's Hospital of Wisconsin will be a prospective, blinded, randomized controlled trial enrolling 20 patients in the pediatric intensive care unit (PICU) with a newly placed central venous catheter (CVC) to receive t-PA or heparin (current standard of care and defined as placebo for this study) to dwell for a minimum of 30 minutes every three days until catheter removal or discharge from the PICU. Primary outcomes would be central line associated blood stream infection (CLABSI) or venous thromboembolism (VTE). Secondary outcomes would be episodes of CVC dysfunction, off study use of t-PA, and bleeding.

Any patient admitted to the PICU and meeting the inclusion criteria will be approached for consent within 72 hours CVC placement. Randomization and administration of study drug/placebo treatment will be initiated within 24 hours of enrollment.

After randomization, study drug/heparin will be infused in the CVC for a dwell duration of 30 minutes-4 hours and then withdrawn (lock therapy) every 3 days until discharge from the PICU, CVC removal or a maximum of 10 doses received. Additional lumens will be treated on subsequent days. Any lumen requiring continuous infusion of vaso-active medication will not receive dwell therapy, evaluated on a day-to-day basis. Timing of instillation of study dwell medication will be adjusted so as not to interfere with medications for patient care.

This single center, pilot study will enroll 20 subjects.

Procedures to be completed for this study are as follows:

After informed consent/assent, the patient will be randomized and assigned to either the treatment arm (t-PA lock) or placebo arm (heparin lock). Randomization will be stratified by age (<5 or ≥5 years old). To maintain the blind, randomization will be done in the investigational pharmacy prior to the dispensing of the study drug/heparin.

Study Treatment and Dosing In subjects randomized to the t-PA, dosing and administration will comply with the Children's Hospital and Health System (CHHS) Policy and Procedure Protocol t-PA Administration for Central Venous Access Devices (CVAD); subjects randomized to the standard of care heparin group will receive an equivalent volume for weight of heparin 10U/ml. The CVC should be flushed with normal saline prior to infusion of study drug/placebo. After dwelling time of 30 minutes-4 hours, study drug/placebo should be withdrawn, check for blood return in CVC and flush line with normal saline as per policy. Each lumen of multi-lumen CVC should be treated every 3 days until patient discharge from PICU, removal of CVC, or a maximum of 10 doses of study drug/placebo are received.

Patient weight Volume Study drug/Placebo 0-10kg 0.5ml 10-20kg 1 ml >20kg 2 ml

These doses by body weight have been approved by the FDA for and CHHS Patient Care Protocol (tPA Administration for Central Venous Access Devices (CVADs) for use in children with CVC and are not associated with significant bleeding. If a 2mg (ml) dose of t-PA is administered by bolus injection directly into the systemic circulation, rather than as a dwell within the CVC, the drug concentration would return to endogenous levels with 30 minutes.

Ultrasound imaging At the end of the study period, a noninvasive ultrasound with doppler will be performed to assess for asymptomatic thrombosis in the blood vessel of the CVC location.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 - ≤ 18 years old
* PICU admission
* CVC placed within 72 hours of enrollment (tunneled such as peripherally inserted central catheter (PICC), Broviac or Hickman, or untunneled) and in place during hospitalization

Exclusion Criteria:

* Pregnancy
* Non-English-speaking subjects and/or parent/guardian
* Platelet count < 20,000
* Active CVC infection-defined as positive blood culture from the in -situ CVC at time of enrollment
* Current radiographically confirmed VTE
* Currently receiving treatment doses of anticoagulation (heparin infusion >15U/kg/hr, enoxaparin injections >=2mg/kg/day or >=60mg/day)
* CVC diameter <1.9 Fr
* Current or previous diagnosis of Heparin Induced Thrombocytopenia or allergy to heparin or t-PA
* Med-a-port catheters

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Alteplase: 10 patients received 30 min-4 hours dwells of alteplase (recombinant t-PA) (2mg/2ml, up to 2mg per dose) to central venous catheter every 3 days (maximum 10 doses)
  alteplase (recombinant t-PA): Medication administered to dwell in central venous catheter
- Heparin: 9 patients received 30 min-4 hours heparin (10U/ml, up to 2 ml per dose) dwells to central venous catheter every 3 days (maximum 10 doses)
  Heparin: Medication administered to dwell in central venous catheter
Period: Overall Study
Arm/Group | Alteplase | Heparin
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — exclusion criteria met | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alteplase | Heparin | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5.5 [1.1 to 11] | 3 [1.25 to 11] | 3 [2 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
CVC type [Count of Participants; unit: Participants]
  Untunneled | 7 | 8 | 15
  PICC | 2 | 1 | 3
  Broviac/Hickman | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Catheter-associated Venous Thrombosis
Description: Catheter-associated Venous Thrombosis upon ICU discharge or 30 days
Time Frame: 30 days or ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Alteplase | Heparin
Number analyzed (Participants) | 10 | 9
Participants | 3 | 3

2. Primary Outcome: Catheter-associated Bloodstream Infection
Description: CLABSI
Time Frame: 30 days or ICU discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Alteplase | Heparin
Number analyzed (Participants) | 10 | 9
Participants | 0 | 0

3. Secondary Outcome: Episodes of CVC Dysfunction
Description: Episodes of CVC dysfunction
Time Frame: 30 days or ICU discharge
Population: episode of CVC dysfunction as inability to flush or draw
Measure: Number; unit: episodes
Arm/Group | Alteplase | Heparin
Number analyzed (Participants) | 10 | 9
episodes | 5 | 2

4. Secondary Outcome: Off Study Use of t-PA
Description: off study use
Time Frame: 30 days or ICU discharge
Population: number of episodes of off-study t-PA use
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Alteplase | Heparin
Number analyzed (Participants) | 10 | 9
doses | 0.5 [0 to 1] | 0 [0 to 0]

5. Secondary Outcome: Clinical Bleeding
Description: clinically significant bleeding
Time Frame: 30 days or ICU discharge
Population: Bleeding events defined as clinically significant
Measure: Number; unit: episodes
Arm/Group | Alteplase | Heparin
Number analyzed (Participants) | 10 | 9
episodes | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days after study completion
Description: clinical bleeding
Arm/Group | Alteplase | Heparin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT03672006/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03672006/ICF_001.pdf